CLINICAL TRIAL: NCT05996315
Title: Ultrasound Guided Supracondylar Nerve Block & Hematoma Block for Closed Reduction of Distal End Radius Fractures - an Observational Study
Brief Title: Ultrasound Guided Supracondylar Nerve Block & Hematoma Block for Closed Reduction of Distal End Radius Fractures
Status: Completed | Type: Observational
Sponsor: Jubilee Mission Medical College and Research Institute (Other)
Responsible Party: Principal Investigator, Dr Roshan Benny, Junior Resident, Jubilee Mission Medical College and Research Institute
Other Study IDs: 40/22/IEC/JMMC&RI
Record Dates: First submitted 2023-05-20; First posted 2023-08-18 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Adults >18 Years With Distal End Radius Fracture Requiring Closed Reduction in Emergency Department
Keywords: distal end radius fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults >18 years with distal end radius fracture: Adults > 18 years with distal end radius fracture requiring closed reduction in Emergency Department
  Interventions: Other: Hematoma block; Other: Supracondylar radial nerve block

INTERVENTIONS:
Other: Hematoma block — A patient who presents to the emergency department with a suspected distal end radius fracture , will be sent for an x-ray. If the X ray-shows a distal end radius fracture a decision to give hematoma block will be taken as per the choice of the treating physician. Patients who do not meet the exclusion criteria are excluded from the study at this phase.
Other: Supracondylar radial nerve block — A patient who presents to the emergency department with a suspected distal end radius fracture will be assessed with a baseline NRS score1 and given analgesics if needed. Further they will be sent for an x-ray. If the X ray-shows a distal end radius fracture a decision to give supracondylar radial nerve block will be taken as per the choice of the treating physician. Patients who do not meet the exclusion criteria are excluded from the study at this phase.

SUMMARY:
Comparison of analgesia between ultrasound guided supracondylar radial nerve block and hematoma block for closed reduction of distal end radius fractures- an observational study

DETAILED DESCRIPTION:
A patient who presents to the emergency department with a suspected distal end radius fracture will be assessed with a baseline NRS score1 and given analgesics if needed. Further they will be sent for an x-ray. If the X ray-shows a distal end radius fracture a decision to give hematoma block or supracondylar radial nerve block will be taken as per the choice of the treating physician. Patients who do not meet the exclusion criteria are excluded from the study at this phase. NRS score 2 is assessed once again prior to block and a Hematoma block/ Supracondylar radial nerve block is given. Needle in and out time will be noted and the pain during needling is evaluated using the NRS score 3. Pain score will further be evaluated for every 10 mins after needle out time for a maximum of 30 mins or when the patient gets adequate analgesia ( NRS score 4a, 4b, 4c, 4d).

If the block is successful, the treating physician will proceed to fracture reduction. If the block is a failure the physician will go for a rescue analgesia. NRS score5 will be evaluated at this stage. Further a NRS score 6 will be assessed 15 minutes post reduction. An x-ray will be checked for the evaluation of the reduction procedure performed and the patient will be discharged or admitted as necessary. The patient will be further followed after 1 week for delayed complications.

ELIGIBILITY:
Inclusion Criteria:

1. Adults > 18 years with distal end radius fracture requiring closed reduction in Emergency Department
2. Patient who legally consent for study

Exclusion Criteria:

1. History of allergy to local anesthetics
2. Pregnant or lactating women
3. Infection or burn with local anaesthetic at injection site
4. Patients having other fractures or significant injuries that are causing pain
5. Patients with hemodynamic instability which includes patients with GCS score less than 15 under influence of alcohol/ inebriated state.
6. Patients on anticoagulants
7. Patients with compromised neurovascular system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who present with isolated distal end radius fracture.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
To compare analgesic effect of supracondylar radial nerve block with hematoma block under ultrasound guidance in closed reduction of distal end radius fractures in emergency department assessed using numerical rating scale. | 60 minute
  To assess the difference in analgesic effect of supracondylar radial nerve block with hematoma block under ultrasound guidance in closed reduction of distal end radius fractures in emergency department assessed using numerical rating scale.

SECONDARY OUTCOMES:
To compare time taken for performing hematoma block & supracondylar radial nerve block | 60minute
  To compare the time taken for hematoma block & supracondylar radial nerve block for closed reduction of distal end radius fracture. Time is noted from needle in to needle out for both technique.
To compare time taken for analgesic effect of hematoma block & supracondylar radial nerve block for closed reduction of distal end radius fracture | 60minute
  compare the analgesic effects of both technique ,which reduces the pain score more during the closed reduction
To compare complication rates of hematoma block & supracondylar radial nerve block for closed reduction of distal end radius fracture | 18months
  Compare the immediate & delayed complications upto 7 days after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency Medicine Department of Jubilee Mission Medical College & Research Institute, Thrissur, Thrissur, Kerala, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maleitzke T, Plachel F, Fleckenstein FN, Wichlas F, Tsitsilonis S. Haematoma block: a safe method for pre-surgical reduction of distal radius fractures. J Orthop Surg Res. 2020 Aug 26;15(1):351. doi: 10.1186/s13018-020-01819-y. PMID 32843043
- [Background] Unluer EE, Karagoz A, Unluer S, Kosargelir M, Kizilkaya M, Alimoglu O, Akoglu H, Aslan C. Ultrasound-guided supracondylar radial nerve block for Colles Fractures in the ED. Am J Emerg Med. 2016 Aug;34(8):1718-20. doi: 10.1016/j.ajem.2016.06.007. Epub 2016 Jun 8. No abstract available. PMID 27342965
- [Background] Tabrizi A, Mirza Tolouei F, Hassani E, Taleb H, Elmi A. Hematoma Block Versus General Anesthesia in Distal Radius Fractures in Patients Over 60 Years in Trauma Emergency. Anesth Pain Med. 2016 Nov 27;7(1):e40619. doi: 10.5812/aapm.40619. eCollection 2017 Feb. PMID 28920036
- [Background] Fathi M, Moezzi M, Abbasi S, Farsi D, Zare MA, Hafezimoghadam P. Ultrasound-guided hematoma block in distal radial fracture reduction: a randomised clinical trial. Emerg Med J. 2015 Jun;32(6):474-7. doi: 10.1136/emermed-2013-202485. Epub 2014 Jul 12. PMID 25016389
- See also: Ultrasound guided haematoma block may be a safe and effective alternative to procedural sedation and analgesia. — https://emj.bmj.com/content/32/6/474
- See also: ultrasound guided radial nerve block is safe — https://pubmed.ncbi.nlm.nih.gov/27342965/